CLINICAL TRIAL: NCT05311228
Title: The Efect of Azithromicyn on Bronchopulmonary Displasia in Extremely Preterm and Very Preterm Infant
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Besse Sarmila, dr. Besse Sarmila, Sp.A, trainee subspecialist neonatology division, principle investigator, clinicalpediatrician, Indonesia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 21050544
Record Dates: First submitted 2022-01-22; First posted 2022-04-05 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Bronchopulmonary Dysplasia; Intraventricular Hemorrhage; Necrotizing Enterocolitis
MeSH Terms: conditions — Bronchopulmonary Dysplasia; Enterocolitis, Necrotizing

STUDY DESIGN:
Intervention Model Description: Two groups, one group intervention and one group control
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Intervention group will give azithromycin for 14 days, 7 days 10 mg/body weight/24 hours, 7 days 5 mg/bw/hours
  Interventions: Drug: Azithromycin Powder
- Control group (No Intervention): No intervention

INTERVENTIONS:
Drug: Azithromycin Powder — Azithromicyn intravena for 14 days
  Arms: Intervention group

SUMMARY:
This study was to see the effectiveness of azithromycin in preventing the incidence of bronchopulmonary dysphasia in extremely preterm and very premature infants. Inclusion criteria were infants with a gestational age of 25-31 weeks 6 days who experienced respiratory distress and their families had agreed to participate in the study, then randomized. The intervention was in the form of giving azithromycin in the intervention group and no intervention was carried out in the control group and then followed up to 36 weeks PMA

ELIGIBILITY:
Inclusion Criteria:

* premature infant 25-31 weeks 6 days with respiratory distress,

Exclusion Criteria:

* multiple congenital anomaly

Ages: 25 Weeks to 32 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes
Enrollment: 120 (Actual)
Dates: Start 2021-06-08 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Bronchopulmonaty Dysplasia | BPD mild room air until 36 weeks PMA, BPD moderate use of oxygen <30% until 36 weeks PMA, BPD severe use of oxygen >30% until 36 weeks PMA
  Use of oxygen suplemantation at least 28 days until 36 weeks PMA

SECONDARY OUTCOMES:
Intraventricular hemorrhage | 1 days-7 days, and 6 weeks
  Sign of IVH from head ultrasonography from USG we can found the sign of IVH grade 1 if we perform head USG and we found bleeding in germinal matriks grade 2 if we perform head USG and we found bleeding intaventricular without ventricle dilatation grade 3 if we perform head USG we found bleeding intraventrucular with dilatation of ventricle grade 4 if we perform head USG and we found bleeding in parenchime
  Head USG perform at 1-7 days and then in 6 weeks
Necrotizing Enterocolitis | 1 days-36 weeks PMA
  Sign and symptoms of NEC from clinical, laboratory, and radiology
  If we found :
  From clinical sign : temperature < 36.5 degree C or > 37.5 degree C, Respiratory rate > 60/min with retraction, abdominal distention Laboratory examination : trombocyte < 100.000/mm3, natrium <135 meq/L, pH < 7.1, BE > -12, CRP > 5 IU Radiology examination : sign of pneumatosis intestinalis
  NEC : clinically + laboratory + radiology

CONTACTS AND LOCATIONS:
Locations (1):
- University of Indonesia, Jakarta, DKI Jakarta, Indonesia

IPD SHARING:
Plan to Share IPD: Undecided
Maybe i will share IPD with other researcher